CLINICAL TRIAL: NCT01284829
Title: Performance of 18F-Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) in the Diagnosis of Indeterminate Adrenal Tumors on Conventional Imaging: A French Prospective Multicentric Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A00705-34; 2010 08 (Other: AP HM)
Record Dates: First submitted 2011-01-13; First posted 2011-01-27 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Adrenal Tumors
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adrenal tumors (Experimental): adrenal tumors
  Interventions: Other: FDG-PET scan

INTERVENTIONS:
Other: FDG-PET scan

SUMMARY:
This is a prospective study which aims to validate a new diagnostic approach in the tissue characterization of adrenal tumors indeterminate on conventional imaging. For this purpose, it is not necessary to have a control group since the diagnostic accuracy in a well defined subset of patients.

Visit 0 : Enrollment, eligibility. Visit 1 : FDG-PET. Visit 2 : Postoperative visit. Visit 3 : 6 months post-PET. Visit 4 : 12 months post-PET.

DETAILED DESCRIPTION:
Primary objective The primary objective is to assess the diagnostic accuracy of FDG-PET, particularly the SUVmax tumor/liver ratio, in the diagnosis of indeterminate adrenal tumors on conventional imaging.

Secondary objectives

* To assess the diagnostic accuracy of the tumor SUVmax, and SUVmax of the tumor/mean SUV of the liver.
* To evaluate the relationship between SUVmax tumor/liver ratio and Weiss score.
* To evaluate the impact of the use of FDG-PET on the treatment options.
* To evaluate the economic impact of FDG-PET in the management of indeterminate adrenal tumors (ancillary study).

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 yrs, male or female;
* Indeterminate adrenal tumor (6.3.1.). The CT must include the calculation of SD and contrast washout and should have been performed within the 30 days before the inclusion visit (visit 0) ;
* Patient insured with public health care system ;
* Patient who accept to participate to the study and to sign the consent document form.

Exclusion Criteria:

* Technical inability to perform FDG-PET.
* Patient's death before final diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-02-04 (Actual); Primary Completion 2013-10-10 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of FDG-PETparticularly the SUVmax tumor/liver ratio, in the diagnosis of indeterminate adrenal tumors on conventional imaging. | 3 YEARS

SECONDARY OUTCOMES:
assess the diagnostic accuracy of the tumorSUVmax, and SUVmax of the tumor/mean SUV of the liver. | 3 YEARS
To evaluate the relationship between SUVmax tumor/liver ratio and Weiss score | 3 years
To evaluate the impact of the use of FDG-PET on the treatment options | 3 years
To evaluate the economic impact of FDG-PET in the management of indeterminate adrenal tumors (ancillary study). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: DAVID TAEB, Principal Investigator — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Guerin C, Pattou F, Brunaud L, Lifante JC, Mirallie E, Haissaguerre M, Huglo D, Olivier P, Houzard C, Ansquer C, Hindie E, Loundou A, Archange C, Tabarin A, Sebag F, Baumstarck K, Taieb D. Performance of 18F-FDG PET/CT in the Characterization of Adrenal Masses in Noncancer Patients: A Prospective Study. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2465-2472. doi: 10.1210/jc.2017-00254. PMID 28431167